CLINICAL TRIAL: NCT02534779
Title: Assessing the Disintegration, Safety, and Acceptability of Placebo Vaginal Inserts for the Delivery of Vaginal Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CONRAD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: D15-134
Record Dates: First submitted 2015-08-21; First posted 2015-08-28 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-06

CONDITIONS: Vaginal Diseases
MeSH Terms: conditions — Vaginal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo Vaginal Insert (Experimental): Placebo insert
  Interventions: Other: Placebo Vaginal Insert

INTERVENTIONS:
Other: Placebo Vaginal Insert — Placebo insert

SUMMARY:
This open-label study will examine the disintegration/disappearance time, safety, and acceptability of placebo vaginal inserts. Participants will use a placebo vaginal insert twice: first for an in-clinic disintegration/safety assessment, and a second time for an at-home acceptability assessment, with safety assessed at the following clinic visit.

DETAILED DESCRIPTION:
This open-label study will examine the disintegration/disappearance time, safety, and acceptability of placebo vaginal inserts. Participants will use a placebo vaginal insert twice: first for an in-clinic disintegration/safety assessment, and a second time for an at-home acceptability assessment, with safety assessed at the following clinic visit.

Participants will be assigned to test their insert during either the follicular or luteal phase of their menstrual cycle, such that the number of women who test it in the follicular phase is approximately equal to the number who test it in the luteal phase.

Once eligibility has been confirmed, the participant will complete an in-clinic disintegration test to estimate the amount of time required for disintegration and complete disappearance of the vaginal insert. Prior to and following the disintegration test, the participant will have a pelvic exam and vaginal swab(s) will be collected for development of adherence measures. Safety will be assessed by naked eye exam and report of adverse events (AEs).

24 to 72 hours following the in-clinic disintegration test, the participant will use the vaginal insert at home and complete a standardized acceptability questionnaire 4 hours and 24 hours after placement. The acceptability questionnaire will be returned to the clinic at the participant's next visit. The final clinic visit will be scheduled 24-72 hours after placement of the vaginal insert used at home.

The final study visit will include a pelvic exam to assess safety and vaginal swab(s) will be collected for development of adherence measures. The participant will exit the study following the final study visit.

This study is designed to test a single placebo vaginal insert, but it is possible additional inserts may become available for testing. Participants may re-enroll in the study for the testing of additional vaginal inserts as they become available.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years, inclusive
* General good health (by volunteer history and investigator judgment)
* Currently having regular menstrual cycles of 21 - 35 days by volunteer report
* Protected from pregnancy, meaning one of the following: Sexually abstinent and planning to remain abstinent for the duration of the study; In a monogamous heterosexual relationship for at least four months with a partner who is not known to be HIV positive and has no known risks for sexually transmitted infections (STIs) and: Couple is using condoms and is willing to use non-spermicidally lubricated condoms throughout the study or One partner is sterilized; or in a monogamous same-sex relationship for at least four months with a partner who is not known to be HIV positive and has no known risks for STIs.
* Willing to abstain from vaginal activity and vaginal product use as required in the protocol
* Vaginal and cervical anatomy that, in the opinion of the investigator, lends itself to easy examination
* Willing to give voluntary consent, sign an informed consent form and comply with study procedures as required by the protocol

Exclusion Criteria:

* History of hysterectomy
* Currently pregnant or within two calendar months from the last pregnancy outcome. Note: If recently pregnant must have had at least two spontaneous menses since pregnancy outcome
* Use of any hormonal contraceptive method in the last 30 days (oral, transdermal, transvaginal, implant, or hormonal intrauterine contraceptive device)
* Injection of Depo-Provera in the last 6 months
* Current use of copper intrauterine device (IUD)
* Currently breastfeeding or having breastfed an infant in the last two months, or planning to breastfeed during the course of the study
* History of sensitivity/allergy to any component of the study products
* Symptomatic reproductive tract infection (RTI)
* Chronic or acute vulvar or vaginal symptoms (pain, irritation, spotting, etc.)
* Known current drug or alcohol abuse which could impact study compliance
* Participation in any other investigational trial (device, drug, or vaginal trial) within the last 30 days or planned participation in any other investigational trial during the study
* History of gynecological procedures (including genital piercing) on the external genitalia, vagina or cervix within the last 14 days
* Abnormal finding on physical examination or a social or medical condition which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Time to disintegration (insert no longer coherent but residual product is visible) | Up to 90 minutes post-insertion
Percent of inserts that partially/fully disintegrate and completely disappear at each time point of observation | Up to 90 minutes post use
Time to complete disappearance | Up to 90 minutes post-insertion

SECONDARY OUTCOMES:
Abnormal findings related to study product on pelvic examination by naked eye exam | Up to 90 minutes post use; 24-72 hours post at-home use
Genitourinary adverse events after use of inserts | Up to 90 minutes post use; 24-72 hours post at-home use

OTHER OUTCOMES:
Responses on acceptability questionnaire after a single use of a vaginal insert | 4 hours and 24 hours post at-home use

CONTACTS AND LOCATIONS:
Overall Officials: Jill Schwartz, MD, Study Chair — CONRAD
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided